CLINICAL TRIAL: NCT05957276
Title: Global Patient Registry of Inherited Retinal Disease
Brief Title: Global Patient Registry of Inherited Retinal Diseases
Acronym: EYERD Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109326; NOPRODRPG0002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2023-06-29; First posted 2023-07-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inherited Retinal Diseases
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Inherited Retinal Diseases (IRDs): Adult and pediatric (greater than or equal to [>=] 3 years) participants with a documented genetic diagnosis of X-linked retinitis pigmentosa (XLRP) or Achromatopsia (ACHM) and any signs or symptoms of IRD or documented retinal changes detected by imaging or electrophysiology.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Standard of Care — Participants will not receive any intervention in this study. Participants will receive standard of care therapy.

SUMMARY:
The purpose of this study is to better understand the natural history of Inherited Retinal Disease (IRD) and help inform patient management.

ELIGIBILITY:
Inclusion Criteria:

For Participant Selection:

* Participant has any clinically documented sign(s) and/or symptom(s) consistent with an Inherited Retinal Disease (IRD), or asymptomatic with documented retinal changes detected by imaging or electrophysiology
* Participant has documented genetic variant(s) (known pathogenic, likely pathogenic, or variants of uncertain significance) in relevant genes for any of the following IRDs: X-Linked Retinitis Pigmentosa (XLRP) and/or Achromatopsia (ACHM)
* Participant or legally acceptable representative has provided informed consent (and participant assent, when applicable) in accordance with local requirements
* Participant is able to have relevant visual and/or retinal assessments performed

For Caregiver Selection:

* Caregiver has consent from the associated participant to participate in the study, or participant assent and consent from their legally acceptable representative
* Male or female aged greater than or equal to (>=)18 years
* Identified by an enrolled participant (or their legally acceptable representative*) as a primary caregiver
* Caregiver has provided informed consent in accordance with local requirements

Exclusion Criteria:

For Participant Selection:

- Participant has received a treatment in an IRD-related interventional trial, or is being screened for an IRD-related interventional trial

For Caregiver Selection:

- Caregiver has an IRD diagnosis and presents with symptoms (visual impairment)

Min Age: 3 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes adult and pediatric participants with a documented genetic diagnosis of XLRP or ACHM and any signs or symptoms of disease.
Sampling Method: Non-Probability Sample
Enrollment: 891 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-07-03 (Estimated); Study Completion 2026-07-03 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity (VA) | Baseline up to 8 years
  VA is a measure of the sharpness of vision. The test uses a chart with letters or symbols of different sizes, at a specific distance, and is reported using various scales, such as fraction, decimal, minimum angle of resolution (MAR), logMAR. When a participant is unable to read a chart, visual acuity can be measured by counting fingers, hand motion, or light perception.
Visual Field (VF) | Baseline up to 8 years
  VF is used to determine scope of vision, including central and peripheral vision. It can determine place, size, and shape of scotoma in vision.

SECONDARY OUTCOMES:
Association Between Inherited Retinal Disease (IRD) Genotype and Visual Acuity | Baseline up to 8 years
  Association between IRD genotype and visual acuity will be reported as incidence of visual acuity for given IRD genotype.
Association Between IRD Genotype and Visual Field | Baseline up to 8 years
  Association between IRD genotype and visual field will be reported as incidence of visual field for given IRD genotype.
Association Between IRD Genotype and Change in Visual Acuity | Baseline up to 8 years
  Association between IRD genotype and change in visual acuity will be reported as change in visual acuity for given IRD genotype.
Association Between IRD Genotype and Change in Visual Field | Baseline up to 8 years
  Association between IRD genotype and change in visual field will be reported as change in visual field for given IRD genotype.
Family History and Inheritance Pattern | Baseline up to 8 years
  Number and relationship with family members diagnosed with IRD will be described.
IRD Variants and Subtypes | Baseline up to 8 years
  Number and distribution of IRD variants and subtypes will be described.
Demographic Characteristics of Participants: Age | Baseline
  Demographic characteristics of participants (age) will be reported.
Demographic Characteristics of Participants: Sex | Baseline
  Demographic characteristics of participants (sex) will be reported.
Demographic Characteristics of Participants: Race | Baseline
  Demographic characteristics of participants (race) will be reported.
Number of Participants With Comorbidities | Baseline
  Number of participants with comorbidities will be reported.
Number of Participants With Various Signs and Symptoms | Baseline
  Number of participants with various signs and symptoms (for example: amblyopia, blindness, corneal disease/dystrophy) will be reported.
Number of Participants With Other Ocular Events | Baseline up to 8 years
  Number of participants with other ocular events will be reported. Other ocular events of interest including cystoid macular edema, macular hole, epiretinal membrane formation, intraocular inflammation, cataracts, glaucoma, chorioretinal atrophy will be described.
Number and Type of Healthcare Professional Visits Prior to Confirmed IRD Diagnosis | Baseline up to 8 years
  Participant diagnostic pathway prior to diagnosis including number and type of healthcare professional visits will be described.
Number and Type of Hospital/Clinic Visit After IRD Diagnosis | Baseline up to 8 years
  Participant management after diagnosis including number and type of hospital/clinic visit will be described.
Medical Resource Utilization | Baseline up to 8 years
  Number and type of hospital/clinic visit, use of assistive device, supportive care, adaptation, and service will be described.
Clinician Global Impression of Severity (CGIS) | Baseline up to 8 years
  CGIS score will be reported for participants with X-linked retinitis pigmentosa (XLRP) and achromatopsia (ACHM) separately. CGIS is a generic, global, 5-point clinician-administered (observer-rated) scale that assesses illness severity. The score ranging from 1 (no symptoms) through 5 (very severe) to assess disease severity. A higher score indicates more severe disease.
Clinical Global Impression of Change (CGIC) | First post-baseline visit up to 8 years
  CGIC score will be reported for XLRP participants. CGIC is a global, generic, 7-point clinician-administered (observer-rated) scale that assesses change in illness severity. The score ranging from 1 (very much improved) through 7 (very much worse). A higher score indicates worsening of disease.
Participant Global Impression of Severity (PGIS) | Baseline up to 8 years
  The PGIS is a 5-point scale to assess disease severity, for participants with XLRP and ACHM separately. The XLRP PGIS measures participant reported disease severity and impact of XLRP on daily activities, items include: daily activities, mobility, mobility under low luminance/at night, and global rating of severity. A higher score indicates more severe disease. The ACHM PGIS measures participant reported disease severity and impact of ACHM on daily activities, items include: photo aversion (indoors and outdoors), impact on daily activities, and global rating of severity. A higher score indicates more severe disease.
Participant Global Impression of Change (PGIC) | First post-baseline visit up to 8 years
  PGIC is a 5-point scale to assess the patient-reported change in disease severity. The XLRP PGIC assesses participant reported perceived change in disease severity and impact of XLRP on daily activities, items include: daily activities, mobility, mobility under low luminance/at night, and global rating of change in severity. A higher score indicates worsening of disease.
Modified Low Luminance Questionnaire (mLLQ) | Baseline up to 8 years
  The mLLQ is a modified version of the original low luminance questionnaire developed for use in eye diseases to assess self-reported task difficulty under low luminance and at night. The mLLQ uses 5-point or 6-point Likert scales, consists of 6 domains: driving, extreme lighting, mobility, emotional distress, general dim lighting, and peripheral vision. There are 3 age versions: the adult (greater than or equal to [>=] 18 years) version includes 30 items, the adolescent (12-17 years) version includes 22 items, and the caregiver (3-11 years) version includes 19 items. Each domain has a score range of 0-100, with higher scores reflecting a higher level of functioning. Scores will be described per age class separately only for participants with XLRP.
Achromatopsia (ACHM) Vision Impact Questionnaire (AVIQ) | Baseline up to 8 years
  The AVIQ was developed to assess the impact of ACHM on functional vision in children and adults. The AVIQ uses 5-point or 6-point Likert scales. There are 3 age versions: the adult/adolescent (>= 12 years) version includes 15 items, the child (8-11 years) version includes 8 items, and the caregiver (5-7 years) version includes 5 items. Scores will be described per age class separately.
Achromatopsia (ACHM) Symptom and Impact Diary | Baseline up to 8 years
  The ACHM symptom and impact diary assesses the severity of key symptoms of photosensitivity and impaired visual acuity, contrast sensitivity, and color vision. There are 3 age versions: the adult/adolescent (>=12 years) version includes 9 items, the child (8-11 years) version includes 9 items, and the caregiver (5-7 years) version includes 16 items. Scores will be described per age class separately.
Hospital Anxiety and Depression Scale (HADS) | Baseline up to 8 years
  The HADS is a 14-item questionnaire to assess the presence of anxiety and depression in individuals aged 16-65 years, using 4-point Likert scales. Summary scores are reported for the 2 domains. Each domain has a score range of 0-21, with higher scores reflecting increased anxiety or depression.
Work Productivity and Activity Impairment (WPAI) | Baseline up to 8 years
  The WPAI is a 6-item questionnaire that measures the effects of IRD symptoms on work productivity and absenteeism and activity impairment outside of work, using dichotomous (Yes/No) and 0-10 numerical rating scale. The productivity loss would be the total work impairment; the sum of absenteeism and presenteeism. Scores are expressed as impairment percentages, with higher scores reflecting more impairment. This questionnaire will be answered by both study participants and caregiver participants.
Caregiver Burden Score | Baseline up to 8 years
  The caregiver burden score is a 14-item questionnaire developed to assess the impact of IRDs on caregivers of children (ages 3-17 years) with an IRD diagnosis, using 4-point or 6-point Likert scales. It measures caregiver burden in terms of perception of their physical and emotional health, relationships, social life, work, and finances. This questionnaire applies to caregivers of minors only.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (75):
- United States (18):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of Southern California, Los Angeles, California
  - UCSF, San Francisco, California
  - Bascom Palmer Eye Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - Ochsner Medical Center, New Orleans, Louisiana
  - John Hopkins Hospital, Baltimore, Maryland
  - Univ of Michigan Medical Center, Ann Arbor, Michigan
  - University Of Minnesota Medical Center, Minneapolis, Minnesota
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - UPMC, Pittsburgh, Pennsylvania
  - Retina Consultants of Texas, Bellaire, Texas
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Houston, Houston, Texas
- Australia (3):
  - Centre for Eye Research Australia, East Melbourne
  - Lions Eye Institute, Nedlands
  - Sydney Children's Hospital, Westmead
- Austria (2):
  - Kepler Universitatsklinikum GmbH, Linz
  - Medizinische Universitaet Wien, Vienna
- Ghent University Hospital, Ghent, Belgium
- Brazil (4):
  - INRET Clínica e Centro de Pesquisa, Belo Horizonte
  - On Oftalmologia LTDA, Pinheiros
  - Clinica Oftalmologica Sao Lucas, São Paulo
  - Instituto De Genetica Ocular, São Paulo
- Sunnybrook Health Sciences Center, Toronto, Ontario, Canada
- China (8):
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital CMU, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Sun YatSen University, Zhongshan Ophthalmic Center, Guangzhou
  - Eye and ENT Hospital of Fudan University, Shanghai
  - Shanghai General Hospital, Shanghai
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Aier Eye Hospital, Shanghai
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark
- Helsingin Yliopistollinen Keskussairaala, Helsinki, Finland
- France (5):
  - CHU Montpellier, Montpellier
  - CHU Nantes, Nantes
  - Centre Hospitalier National d'Ophtalmologie des Quinze-Vingts, Paris
  - Hôpital Necker-Enfants Malades, Paris
  - Hopitaux universitaires de Strasbourg, Srasbourg
- Universitatsklinikum Bonn, Bonn, Germany
- Israel (2):
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Arcispedale S. Anna Ferrara, Ferrara
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Ospedale San Raffaele, Milan
  - ASST Santi Paolo e Carlo, Milan
  - Azienda Ospedaliera Univ.- Università Degli studi della Campania - Luigi Vanvitelli, Napoli
  - Policlinico Universitario Agostino Gemelli, Roma
  - IRCCS Fondazione G.B. Bietti per lo Studio e la Ricerca in Oftalmologia ONLUS, Roma
- Japan (4):
  - Kyushu University Hospital, Fukuoka
  - National Hospital Organization Tokyo Medical Center, Meguro-ku
  - Nagoya University Hospital, Nagoya
  - Mie University Hospital, Tsu
- South Korea (3):
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (6):
  - Hosp. Univ. de Bellvitge, Barcelona
  - Hosp. Sant Joan de Deu, Barcelona
  - Hosp. Univ. Donostia, Donostia / San Sebastian
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Virgen Macarena, Seville
- Switzerland (2):
  - University Hospital Basel, Eye Clinic/Institute of Molecular and Clinical, Basel
  - Universite de Lausanne, Hopital ophtalmique Jules-Gonin, Lausanne
- United Kingdom (6):
  - University Hospital Wales, Cardiff
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Sunderland Eye Infirmary, Sunderland

IPD SHARING:
Plan to Share IPD: No